CLINICAL TRIAL: NCT05041231
Title: Effects of Using Custom Photobiomodulation Therapy for the Treatment of Osteoarthritis of the Fingers and Rhizarthrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vita Care (Other)
Collaborators: Tegos S.A. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 133
Record Dates: First submitted 2021-08-25; First posted 2021-09-10 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Osteoarthritis; Osteoarthritis Finger; Osteoarthritis Hand; Osteoarthritis Both Hands
MeSH Terms: conditions — Osteoarthritis | interventions — Low-Level Light Therapy; Lasers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham (group A) (Sham Comparator): Treatment procedure performed with the device that will not provide the bioactive light (laser)
  Interventions: Device: Sham Photobiomodulation therapy (Sham PBT)
- PBT (group B) (Experimental): Treatment procedure performed with the device that will provide the bioactive light (laser)
  Interventions: Device: Photobiomodulation therapy (PBT)

INTERVENTIONS:
Device: Photobiomodulation therapy (PBT) — Any invasive procedures will be done. The treatment in question will be done by a device that looks like a bracelet, which is placed on the hand/fingers to emit light/laser and does not cause pain or temperature change. There will be 8 photobiomodulation sessions, 2 per week, 10 minutes each session.
  The dosimetric parameters of the therapy will be carried out in a standardized and personalized way, with programming of the light and all the necessary information so that the device can carry out the application of the treatment application of electromagnetic waves in the red and infrared spectral range 660-1000 nm).
  Other Names: Laser
  Arms: PBT (group B)
Device: Sham Photobiomodulation therapy (Sham PBT) — Similar to active PBT, however, the device will not provide the active electromagnetic waves)
  Other Names: Sham Laser
  Arms: Sham (group A)

SUMMARY:
Osteoarthrosis (OA), a multifactorial degenerative process, is responsible for joint pain and functional limitation. In the hand, more specifically in the proximal and distal interphalangeal joints of the fingers, it is one of the sites of greatest manifestation of the disease. Numerous treatments, whether drug, rehabilitation or surgery, have been proposed with the aim of both interrupting the natural evolution of the disease and alleviating or stopping the symptoms. This study aims to evaluate the effectiveness of personalized Photobiomodulation Therapy (PBT) with regard to alleviating symptoms and improving the quality of life of these patients with the disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological diagnosis of OA of the fingers of the hand and Rizarthrosis
* Patients with pain for at least 3 months
* Patients undergoing treatment and rehabilitation for finger OA and rhizarthrosis
* Patient with good understanding of the Portuguese language who agrees to participate and sign the ICF

Exclusion Criteria:

* Posttraumatic arthritic changes
* Systemic inflammatory arthritis (Rheumatoid Arthritis, Lupus Erythematosus, Psoriasis…)
* Patients with local or systemic, acute or chronic infections

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Pain at | 4 weeks and 2 months
  Visual analogue scale for pain
Change from Baseline Arm, Shoulder and Hand Disability | 4 weeks and 2 months
  The Disabilities of the Arm, Shoulder and Hand Score

SECONDARY OUTCOMES:
Change from Baseline Hand grip | 4 weeks and 2 months
  Hand grip strenght measured by Digital Hand Dynamometer
Change from Baseline Pinch force | 4 weeks and 2 months
  Pulp to pulp (pinch) force
Willingness to recommend the treatment | 4 weeks and 2 months
  Net Promoter Score
Change from Baseline Hand Disability | 4 weeks and 2 months
  Brief Michigan questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mateus Saito, PhD, Principal Investigator — Medical Director Instituto Vita
Locations (1):
- Instituto Vita, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No